CLINICAL TRIAL: NCT04726202
Title: Impact of Semi-automated Proposal and Optimization of Diagnoses and Surgical Procedures for Precoding: a Randomized Controlled Trial
Status: Completed | Type: Observational
Sponsor: Thomas Steffen (Other)
Responsible Party: Sponsor-Investigator, Thomas Steffen, Deputy Head of Department, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Other Study IDs: Chir201902
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Diagnosis-Related Groups; Healthcare Common Procedure Coding System
Keywords: DRG; Diagnosis-Related Groups; ICD; reimbursement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control arm: standard procedure of coding at hospital
  Interventions: Other: Standard procedure
- Precoding arm: Coding of the standard procedure will be reviewed and corrected
  Interventions: Other: precoding

INTERVENTIONS:
Other: Standard procedure — Coding of cases follows the standard procedures established at the hospital
  Groups: Control arm
Other: precoding — Standard coding will be reviewed by dedicated physicians and corrected or extended if necessary.
  Coding will compared to the written OP report for consistency. Dedicated physician visits patients daily (in addition to routine visits). Dedicated physicians review discharge report and will make changes and additions. DRG coding will be adapted to results from visits and discharge report.
  Groups: Precoding arm

SUMMARY:
The hypothesis of present study is that the daily monitoring and optimization of DRG coding is associated with higher reimbursement. Therefore, the primary objective is to determine if the daily monitoring and optimization of DRG coding of individual cases leads to better proceeds per day.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing surgery as inpatients (at least one night stay)
* treated at the Kantonsspital St. Gallen, St. Gallen site

Exclusion Criteria:

* surgery as outpatients
* surgery at the Rorschach and Flawil sites
* patients operated on by the Department of Surgery, but hospitalized at another department of the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing inpatient surgery in the fields of General, Visceral, Endocrine or Transplantation Surgery
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
reimbursement per day at hospital | 8 months
  total reimbursement per arm divided by the total stay of the patients in the arm in days

SECONDARY OUTCOMES:
Length of hospital stay | 8 months
  length of hopital stay in full days including entry and discharge day
Total reimbursement per case | 8 months
  reimbursement in Swiss Francs per case
case mix index per case | 8 months
  Financial department will provide the cost weight/case mix index per case
Severity of perioperative complications | 8 months
  complications during hospitalisation will be graded according to the Clavian-Dindo scale. In case of multiple complications the highest grade will be taken.
readmission rate | 8 months
  Rate of case related readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Steffen, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Department of Surgery, Cantonal Hospital of St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fillit H, Geldmacher DS, Welter RT, Maslow K, Fraser M. Optimizing coding and reimbursement to improve management of Alzheimer's disease and related dementias. J Am Geriatr Soc. 2002 Nov;50(11):1871-8. doi: 10.1046/j.1532-5415.2002.50519.x. PMID 12410910
- [Background] Fetter RB, Freeman JL. Diagnosis related groups: product line management within hospitals. Acad Manage Rev. 1986 Jan;11(1):41-54. PMID 10311457
- [Background] Fetter RB. Hospital payment based on diagnosis-related groups. J Soc Health Syst. 1992;3(4):4-15. PMID 1288673
- [Background] Freeman JL, Fetter RB, Park H, Schneider KC, Lichtenstein JL, Hughes JS, Bauman WA, Duncan CC, Freeman DH Jr, Palmer GR. Diagnosis-related group refinement with diagnosis- and procedure-specific comorbidities and complications. Med Care. 1995 Aug;33(8):806-27. doi: 10.1097/00005650-199508000-00006. PMID 7637403
- [Background] Hughes JS, Lichtenstein J, Fetter RB. Procedure codes: potential modifiers of diagnosis-related groups. Health Care Financ Rev. 1990 Fall;12(1):39-46. PMID 10113461
- [Background] Geuss S, Jungmeister A, Baumgart A, Seelos R, Ockert S. [Prospective DRG coding : Improvement in cost-effectiveness and documentation quality of in-patient hospital care]. Chirurg. 2018 Feb;89(2):138-145. doi: 10.1007/s00104-017-0555-4. German. PMID 29188352
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- See also: OnlineGrouper — https://grouper.swissdrg.org/swissdrg/single
- See also: Common Terminology Criteria for Adverse Events (CTCAE) — https://www.eortc.be/services/doc/ctc/CTCAE_4.03_2010-06-14_QuickReference_5x7.pdf
- See also: Federal Act on Data Protection (FADP) — https://www.admin.ch/opc/en/classified-compilation/19920153/index.html
- See also: Human Research Act (HRA) — https://www.admin.ch/opc/de/classified-compilation/20061313/index.html
- See also: Ordinance on Clinical Trials in Human Research (ClinO) — https://www.admin.ch/opc/de/classified-compilation/20121176/index.html

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT04726202/Prot_SAP_000.pdf